CLINICAL TRIAL: NCT03355235
Title: Brilliant Study: Assessing Cognition in Myeloma Patients Undergoing Transplant
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00045767; CCCWFU 02117 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2017-10-20; First posted 2017-11-28 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-07

CONDITIONS: Stem Cell Transplant Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cognitive assessment using standardized tools: cognitive assessment using standardized tools pre and post transplant.

SUMMARY:
The overall objectives in this study are to identify patterns of cognitive impairment pre- and post-transplant, to assess the similarities of scores of the three cognitive assessments in myeloma patients who undergo autologous stem cell transplant, and to determine if patients prefer the self-assessment, Self-Administered Gerocognitive Exam (SAGE) or the healthcare applied Montreal Cognitive Assessment (MoCA) assessment.

DETAILED DESCRIPTION:
The overall objectives in this study are to identify patterns of cognitive impairment pre- and post-transplant, to assess the similarities of scores of the three cognitive assessments in myeloma patients who undergo autologous stem cell transplant, and to determine if patients prefer the self-assessment, Self-Administered Gerocognitive Exam (SAGE) or the healthcare applied Montreal Cognitive Assessment (MoCA) assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple myeloma
* Patients who will undergo pre-transplant evaluation with intentions to proceed to autologous stem cell transplant after stem cell collection.
* Patients willing and able to understand and sign an informed consent form
* Patients 18 yrs of age or older

Exclusion Criteria:

* Patients with unstable psychiatric illness within the past 3 months of study enrollment.
* Patients who are considered unable to perform study evaluations at the investigator's discretion.
* Patients who are unable to read. (If patients require reading glasses, they must be worn at time of test.)
* Patients who do not proceed to stem cell transplant within 60 days of stem cell collection will be excluded from study.
* Patients who receive more than one cycle of chemotherapy between the time of stem cell collection and transplant will be excluded from study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 4.2.1 Patients with multiple myeloma being considered for transplant and scheduled to undergo pre-transplant evaluation
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-08-27 (Actual)

PRIMARY OUTCOMES:
Scores of the PROMIS Cognitive Function, short form 8a | Before to approximately 100 days after transplant
  Will be assessed by Patient Reported Outcomes Measurement Information System (PROMIS) Cognitive Function, short form 8a. The mean scores (and standard deviations) for each time points will be presented.
Scores of the Self-Administered Gerocognitive Exam (SAGE) | Before to approximately 100 days after transplant
  Will be assessed by the Self-Administered Gerocognitive Exam (SAGE). The mean scores (and standard deviations) for each time points will be presented.
Scores of the Montreal Cognitive Assessment (MoCA) | Before to approximately 100 days after transplant
  Will be assessed by Montreal Cognitive Assessment (MoCA). The mean scores (and standard deviations) for each time points will be presented.
Changes in scores of the PROMIS Cognitive Function, short form 8a | Before to approximately 100 days after transplant
  Will be assessed by Patient Reported Outcomes Measurement Information System (PROMIS) Cognitive Function, short form 8a. The mean changes in scores will be presented. The difference in each cognitive tests will be evaluated using a paired t-test to determine if any change has occurred.
Changes in scores of the Self-Administered Gerocognitive Exam (SAGE) | Before to approximately 100 days after transplant
  Will be assessed by the Self-Administered Gerocognitive Exam (SAGE). The mean changes in scores will be presented. The difference in each cognitive tests will be evaluated using a paired t-test to determine if any change has occurred.
Changes in scores of the Montreal Cognitive Assessment (MoCA) | Before to approximately 100 days after transplant
  Will be assessed by Montreal Cognitive Assessment (MoCA). The mean changes in scores will be presented. The difference in each cognitive tests will be evaluated using a paired t-test to determine if any change has occurred.

SECONDARY OUTCOMES:
Agreement between cognitive test (PROMIS 8a and SAGE) | Up to approximately 100 days after transplant
  Evaluate how each tests score is in agreement with the other using statistics correlations.examiner-implemented cognitive assessment, MoCA. Will assess the correlation of the tests before and post-transplant as well as the correlation of the change in scores.
Agreement between cognitive test (PROMIS 8a and MoCA) | Up to approximately 100 days after transplant
  Evaluate how each tests score is in agreement with the other using statistics correlations.
Agreement between cognitive test (SAGE and MoCA) | Up to approximately 100 days after transplant
  Evaluate how each tests score is in agreement with the other using statistics correlations.
Patients' preference between self-assessment tools Questionnaire | Up to 1 year
  Will assess the preference between SAGE and examiner-implemented, MoCA using the Assessment Preference questionnaire. Will present the frequency of preference. Will then test if the proportion is equal to 50% or if one of the assessments is significantly preferred over the other.

CONTACTS AND LOCATIONS:
Overall Officials: Cesar Rodriguez, MD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No